CLINICAL TRIAL: NCT06896578
Title: Lateral Lymph Nodes in Rectal Cancer Attitude Study
Brief Title: Latitude - Lateral Lymph Node Attitude Study
Acronym: Latitude
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Latitude
Record Dates: First submitted 2025-01-09; First posted 2025-03-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: Rectal Neoplasm Malignant
Keywords: lateral lymph nodes; Quality of life; local recurrence; thrombosis; lymph oedema; lateral lymph node dissection
MeSH Terms: conditions — Rectal Neoplasms; Thrombosis

STUDY DESIGN:
Intervention Model Description: Patients will be treated according to their findings on primary MRI. They will initiallly be divided into two groups: No neoadjuvant treatment or neoadjuvant treatment. If no neoadjuvant treatment the patients undergo rectal surgery.
  If neoadjuvant treatment and lateral lymph nodes remain after neoadjuvant treatment (size >4 mm) then the patients will undergo lateral lymph node dissection.
  If neoadjuvant treatment and lateral lymph nodes are ≤4 mm after neoadjuvant treatment then the patients will undergo rectal surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectal cancer surgery without lateral lymph node dissection (No Intervention): Rectal cancer surgery without lateral lymph node dissection. Applicable if no lateral lymph nodes on primary MRI or lateral lymph nodes ≤4 mm after neoadjuvant treatment No lateral lymph node dissection
- Rectal cancer surgery with lateral lymph node dissection (Experimental): Rectal cancer surgery with lateral lymph node dissection. Applicable if lateral lymph nodes on primary MRI that persist after neoadjuvant treatment (> 4 mm) .
  Lateral lymph node dissection
  Interventions: Procedure: Lateral lymph node dissection

INTERVENTIONS:
Procedure: Lateral lymph node dissection — Removal of lateral lymph nodes in the obturator and internal iliac compartment including fatty tissue, but excluding vascular and nervous tissue
  Other Names: Lateral lymph node clearance; Lateral lymph node removal
  Arms: Rectal cancer surgery with lateral lymph node dissection

SUMMARY:
Patients with advanced rectal cancer can sometimes have suspected tumour affected lymph nodes outside the standard operating field. These patients often receive preoperative treatment before surgery. There is a lack of consensus on what to do if there is remaining suspicion of tumour affected lymph nodes after the preoperative treatment. Removal of the lymph nodes using a broader surgical field with dissection of the lateral side-wall is often suggested, but the oncologic outcome is uncertain, and so is the patient reported outcome in terms of side effects.

This study aims to study the surgical treatment of tumour affected lateral lymph nodes to understand what lymph nodes require removal, and what effect that will have on oncologic outcome and the patient's function and QoL.

DETAILED DESCRIPTION:
Patients with advanced rectal cancer will receive standard care, if lateral lymph nodes exist after neoadjuvant treatment they will be operated accordingly. The focus will be to compare two groups (with and without lateral lymph node clearance) regarding function, QoL and oncologic outcome.

We will also aim to identify features on MRI to improve diagnostic ability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* written informed consent
* adenocarcinoma verified tumour below ≤ 8 cm from anal verge measured by rectoscopy and/or MRI
* clinical tumor (cT) stage cT3, cT4a or cT4b on MRI or
* adenocarcinoma verified tumour at any height ≤ 15 cm from anal verge measured by rectoscopy and/or MRI regardless of T/N stage with visible lateral lymph node (according to definition 2.4.2) on pre-therapeutic MRI or PET-CT

Exclusion Criteria:

* Not biopsy confirmed rectal cancer (adenocarcinoma)
* Recurrent rectal cancer
* Age below 18
* Participation in other trials in conflict with the protocol and end-points of the Latitude study
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | Three years
  A tumour recurrence within the lesser pelvis, below the level of the promontory. (This does not include carcinomatosis if there are other signs of carcinomatosis in the abdominal cavity). Diagnosis made clinically (radiology) or by pathology

SECONDARY OUTCOMES:
Complications according to a composite outcome | 90 days
  Composite outcome including:
  * Comprehensive Complications index
  * Lymphedema (answer yes to questionnaire regarding swelling in right/left groin or leg)
  * Thrombosis (registration in CRF) and questionnaire
Lateral local recurrence | 3 years
  A tumour recurrence located in the lateral compartments within the lesser pelvis, below the level of the promontory. (This does not include carcinomatosis if there are other signs of carcinomatosis in the abdominal cavity). Diagnosis made clinically (radiology) or by pathology
Lateral local recurrence | 5 years
  A tumour recurrence located in the lateral compartments within the lesser pelvis, below the level of the promontory. (This does not include carcinomatosis if there are other signs of carcinomatosis in the abdominal cavity). Diagnosis made clinically (radiology) or by pathology
Surgical morbidity (including reoperations) (Clavien Dindo score I-V) | 90 days
  Clavien-Dindo IIIb and more measured as proportion
Surgical morbidity measured as Comprehensive Complications index (lower score = less complications) | 90 days
  All complications registered according to Clavien-Dindo using a calculator to identify a combination of the number and the severity of complications.
Perioperative blood loss | 0-24 hours
  Blood loss during the surgical procedure: Registration in operative CRF (ml in suction + estimation by anaesthesiologist)
Total operating time | 0-24 hours
  Registration in operative CRF (op start and op end)
Length of hospital stay | during the first hospitalization until discharge after first surgery, measured within 3 months of the first surgical proceu
  Total days in hospital including referral to other hospital
Total length of hospital stay | 365 days = 1 year
  Total number of days including readmissions
Number of patients with postoperative thrombosis (deep venous thrombosis and/or pulmonary thrombosis) | 1 year
  Clinical or radiological or patient reported thromobsis
Number of patients with postoperative thrombosis (deep venous thrombosis and/or pulmonary thrombosis) | 2 years
  Clinical or radiological or patient reported thromobsis
Number of patients with postoperative thrombosis (deep venous thrombosis and/or pulmonary thrombosis) | 3 years
  Clinical or radiological or patient reported thromobsis
Health related Quality of life | 1 month postop
  Health related QoL, Measured in QoL questionnaire, a likert scale question 1-7 where 7 is the best possible QoL.
Health related Quality of life | 1 year
  Health related QoL, Measured in QoL questionnaire, a likert scale question 1-7 where 7 is the best possible QoL.
Health related Quality of life | 2 years
  Health related QoL, Measured in QoL questionnaire, a likert scale question 1-7 where 7 is the best possible QoL.
Health related Quality of life | 3 years
  Health related QoL, Measured in QoL questionnaire, a likert scale question 1-7 where 7 is the best possible QoL.
Urinary function | 1 month
  Measured in QoL questionnaire focus on incontinence, emptying difficulties and urgency using direct questions, not a score. Clinimetric approach.
Urinary function | 1 year
  Measured in QoL questionnaire focus on incontinence, emptying difficulties and urgency using direct questions, not a score. Clinimetric approach.
Urinary function | 2 years
  Measured in QoL questionnaire focus on incontinence, emptying difficulties and urgency using direct questions, not a score. Clinimetric approach.
Urinary function | 3 years
  Measured in QoL questionnaire focus on incontinence, emptying difficulties and urgency using direct questions, not a score. Clinimetric approach.
Sexual function | 1 year
  Measured in QoL questionnaire, focus on both function and quality using direct questions, not a score. Clinimetric approach.
Sexual function | 2 years
  Measured in QoL questionnaire, focus on both function and quality using direct questions, not a score. Clinimetric approach.
Sexual function | 3 years
  Measured in QoL questionnaire, focus on both function and quality using direct questions, not a score. Clinimetric approach.
Bowel and stoma function | 1 year
  Measured in QoL questionnaire, major LARS (21-42 points)
Bowel and stoma function | 2 years
  Measured in QoL questionnaire, major LARS (21-42 points)
Bowel and stoma function | 3 years
  Measured in QoL questionnaire, major LARS (21-42 points)
Health economic analysis | 1 year
  A total health economic analysis including societal costs
Mortality | 1 year
  Dead by any cause
Mortality | 2 years
  Dead by any cause
Mortality | 3 years
  Dead by any cause
5- year overall survival | 5 years
  Survival at 5 years
Pain according to brief pain inventory | 1 month
  Measured in QoL questionnaire brief pain inventory with four pain severity items and seven pain interference items rated on 0-10 scales, and the question about percentage of pain relief by analgesics
Pain according to brief pain inventory | 1 year
  Measured in QoL questionnaire brief pain inventory with four pain severity items and seven pain interference items rated on 0-10 scales, and the question about percentage of pain relief by analgesics
Pain according to brief pain inventory | 2 years
  Measured in QoL questionnaire brief pain inventory with four pain severity items and seven pain interference items rated on 0-10 scales, and the question about percentage of pain relief by analgesics
Pain according to brief pain inventory | 3 years
  Measured in QoL questionnaire brief pain inventory with four pain severity items and seven pain interference items rated on 0-10 scales, and the question about percentage of pain relief by analgesics
MRI interobserver variability | First month
  Comparing MRI assessment at baseline between different centers to determine specificity and sensitivity of MRI assessment
MRI interobserver variability | First 6 months
  Comparing MRI assessment at baseline between different centers to determine specificity and sensitivity of MRI assessment
MRI vs pathology | First 6 months
  Comparing MRI assessment with pathology report, diagnostic (pretreatment) and post treatment MRI compared with pathology report
ctDNA at diagnosis | Values at diagnosis, perioperatively and post treatment in relation to cancer recurrence
  Value of ctDNA at diagnosis, the possible correlation with malignant lymph nodes
Value of immunoscore to predict response, and presence of lateral lymph nodes | 1 month
  Is high Immunoscore related to malignant lymph nodes? Diagnostic biopsies will be sectioned, stained with immunohistochemistry will be correlated to lymph nodes on MRI
Value of immunoscore to predict response, and presence of lateral lymph nodes | Perioperative biopsies (within 6 weeks from inclusion)
  Is high Immunoscore related to malignant lymph nodes? Diagnostic biopsies will be sectioned, stained with immunohistochemistry will be correlated to lymph nodes on pathology
Evaluation dose/fraction in relation to response to treatment | Within the first 6 months.
  Details from CRF during treatment planning as well as prospectively collected treatment plans
Evaluation of number of fractions n relation to response to treatment | Within the first 6 months
  Details from CRF during treatment planning as well as prospectively collected treatment plans
Evaluation of final dose to tumor and elective LN volume | Within the first 6 months
  Details from CRF during treatment planning as well as prospectively collected treatment plans

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, MD PhD, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No